CLINICAL TRIAL: NCT07244055
Title: Effects Of Animal Fun Program On Motor Skills In Children With Developmental Coordination Disorder
Brief Title: Effects of Animal Fun Program in Children With DCD.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/MAIRA SHAHZAD
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Child Development
Keywords: Animal Fun program; DCD developmental coordination disoder; BOT 2 (Bruininks-Oseretsky Test of Motor Proficiency )
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial investigates the effects of animal fun program on motor skills in children with developmental coordination disorder. The study involves 40 children from normal school age group 6 to 12 year old, who will be randomly assigned to one of the two groups for a six-week intervention period. Key performance outcomes
  -body management truck control, locomotion, balance ,object control,body sequencing social and emotional control will be assessed both before and after the intervention.This study aims to address this gap by evaluating the effects of the Animal Fun Program on both fine and gross motor activity levels in children diagnosed with DCD. By examining objective motor outcomes and child engagement, the study seeks to determine whether this novel, enjoyable intervention can enhance traditional therapy methods, leading to improved motor development and overall quality of life for children with DCD. Data will be analyzed through SPSS version 27.00.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group. The intervention will be the Animal Fun program, (Experimental): The Animal Fun program consists of nine modules: Body Management, Locomotion, Object Control, Body Sequencing, Body and Kinesthetic Management, Fine Motor Planning, Tool Control, Hand Skills, and Social/Emotional Development. 90-minute session , 10 min for each module four days per week, will be preferable for these activities over a 6-week duration
  Interventions: Other: animal fun program
- control group (Other): Children in the controlled group will be engaged in regular playful physical activities, e.g, Ball catch and throw, trampoline jumping, and running, squats etc is recruited to the other group daily.
  Interventions: Other: control group

INTERVENTIONS:
Other: animal fun program — The Animal Fun program consists of nine modules: Body Management, Locomotion, Object Control, Body Sequencing, Body and Kinesthetic Management, Fine Motor Planning, Tool Control, Hand Skills, and Social/Emotional Development will be intervened to students diagnosed with developmental coordination disorder from 6 years to 12 years of age thruogh DCDQ version 7 and results will be evaluated by usuing BOT/2 .
  Arms: Experimental group. The intervention will be the Animal Fun program,
Other: control group — Children will be engaged in daily playful exercises such as running, trampoline jumping,squats ball catch and throw etc.
  Other Names: Daily physical play activities
  Arms: control group

SUMMARY:
This randomized clinical trial investigates the effects of animal fun program on motor skills in children with developmental coordination disorder. The study involves 40 children from normal school age group 6 to 12 year old, who will be randomly assigned to one of the two groups for a six-week intervention period. Key performance outcomes

-body management truck control, locomotion, balance ,object control,body sequencing social and emotional control will be assessed both before and after the intervention.This study aims to address this gap by evaluating the effects of the Animal Fun Program on both fine and gross motor activity levels in children diagnosed with DCD. By examining objective motor outcomes and child engagement, the study seeks to determine whether this novel, enjoyable intervention can enhance traditional therapy methods, leading to improved motor development and overall quality of life for children with DCD. Data will be analyzed through SPSS version 27.00.

DETAILED DESCRIPTION:
This randomized clinical trial investigates the effects of animal fun program on motor skills in children with developmental coordination disorder. The Animal Fun program was designed to enhance the motor ability of young children by imitating the movements of animals in a fun, inclusive setting. The efficacy of this program will be investigated through a randomized controlled trial. Data will be collected from the normal schools The intervention Animal fun program consists of nine modules and will be given thrice a week for forty minutes, whereas the control group includes normal physical activity.. The study will be completed in six weeks after approval of the synopsis. The study will include 40 kids, male and female. Inclusion criteria for the study will include patients diagnosed with DCD through the DCDQ version 7 questionnaire. Data will be collected from children aged 6 to 12 years old. Changes in motor performance were examined using the Bruininks-Oseretsky Test of Motor Proficiency 2 will be collected from different schools with normal population . This program includes nine modules based on body management truck control, locomotion, balance ,object control,body sequencing social and emotional control will be assessed both before and after the intervention.This study aims to address this gap by evaluating the effects of the Animal Fun Program on both fine and gross motor activity levels in children diagnosed with DCD. By examining objective motor outcomes and child engagement, the study seeks to determine whether this novel, enjoyable intervention can enhance traditional therapy methods, leading to improved motor development and overall quality of life for children with DCD.Data will be analyzed through SPSS version 27.0

ELIGIBILITY:
Inclusion Criteria:

* Children with diagnosed with DCD by DCDQ 7 questionnaire
* Not receiving any intervention within the last 6 months
* Mentally stable enough to participate in physical activity

Exclusion Criteria:

* Medical condition contraindicating active movements

  * Intellectual disability.
  * Children with any other syndrome and progressive neurodevelopmental diseases

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
DCDQ'07 | Baseline, 1st week and 6th week
  The Developmental Coordination Disorder Questionnaire 2007 (DCDQ'07) is a questionnaire for parents aiming at identifying subtle motor problems in children aged 8 to 14 years 6 months. The questionnaire consists of 15 items divided into three factors: Control during movement, Fine motor and handwriting, and General coordination. Although the DCDQ'07 is a reliable and valid instrument it cannot by itself be used to identify DCD.

SECONDARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency-version 2 Short Form (BOT-2SF). | Baseline, 1st week and 6th week]]
  ). Motor performance was measured using the BOT-2SF. The long version, described as the most widely used test of motor proficiency it contains 53 items, whereas the short form has 14 items. As the long form takes at least 40- 60 minutes to administer, the short form was chosen for this study,
  given the young 7 age of the children. The long form has excellent test-retest and inter-rater reliability. Although few studies have examined the psychometric properties of the short form, the inter-rater reliability to be greater than 0.90, test-retest reliability was greater than 0.80, and internal consistency as generally acceptable (> .80), although at ages 4 and 8 years, correlations ranged from 60 to .92
  60 to .92
  ). Motor performance was measured using the BOT-2SF. The long version, described as the most widely used test of motor proficiency it contains 53 items, whereas the short form has 14 items. As the long form takes at least 40- 60 minutes to administer, the short form

CONTACTS AND LOCATIONS:
Overall Officials: Maira Shahzad, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum DA. The Cinderella of psychology: the neglect of motor control in the science of mental life and behavior. Am Psychol. 2005 May-Jun;60(4):308-17. doi: 10.1037/0003-066X.60.4.308. PMID 15943523